CLINICAL TRIAL: NCT03422289
Title: Improved Effects of Myo-inositol in Association With Alpha-lactalbumin in PCOS Women
Brief Title: Improved Effects of MI Plus Alpha-LA in PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MI + alpha-LA
Record Dates: First submitted 2018-01-10; First posted 2018-02-05 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Polycystic Ovary Syndrome
Keywords: myo-inositol; alpha-lactalbumin; anovulation; infertility
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anovulation; Infertility | interventions — Inositol; Folic Acid; Lactalbumin

STUDY DESIGN:
Intervention Model Description: All the patients were given orally Inofolic® (Lo.Li. Pharma, Rome, Italy), containing 2 g myo-inositol and 0.2 mg folic acid twice a day for three months, in order to induce ovulation. Then, non-responder partecipants were administered orally with 2 g myo-inositol plus 50 mg α-lactalbumin, twice a day for three months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myo-inositol + folic acid (Experimental): 2 g myo-inositol and 0.2 mg folic acid orally twice a day for three months, in order to induce ovulation.
  Interventions: Dietary Supplement: myo-inositol plus folic acid
- Myo-inositol + folic a. + α-lactalbumin (Experimental): 2 g myo-inositol and 0.2 mg folic acid plus 50 mg α-lactalbumin, twice a day for three months in order to test if α-lactalbumin addition allows to induce ovulation
  Interventions: Dietary Supplement: myo-inositol plus folic acid plus alpha-lactalbumin

INTERVENTIONS:
Dietary Supplement: myo-inositol plus folic acid — this treatment is made in the first phase of the study for three months
  Arms: Myo-inositol + folic acid
Dietary Supplement: myo-inositol plus folic acid plus alpha-lactalbumin — this treatment is made in the second phase of the study and it has a new molecule added to the previous ones administered in the first phase of the study
  Arms: Myo-inositol + folic a. + α-lactalbumin

SUMMARY:
PCOS patients are initially treated with 2 g myo-inositol and 0.2 mg folic acid, two times per day by oral route, for three months. Among them, the subjects who have not ovulated despite this treatment are administered with 2g myo-inositol and 0.2 mg folic acid plus 50 mg α-lactalbumin for three months. Most of them improve and achieve ovulation. Therefore, the combination of α-lactalbumin with myo-inositol allows to get a significant result in the treatment of PCOS patients.

DETAILED DESCRIPTION:
Polycystic ovary syndrome is a complex chronic condition inducing several related disorders, such as subfertility and pregnancy complications. So far myo-inositol, successfully used in PCOS, has not been always effective in all patients. Aiming at overcoming this drawback, we tested a new formulation with myo-inositol and α-lactalbumin, in consideration of the effects exerted by α-lactalbumin in favoring molecule passage among body compartments, and also in consideration of its anti-inflammatory activity.

Only PCOS patients, according to Rotterdam ESHRE-ASRM criteria, with anovulation and infertility > 1 year, were included in the study. Following a treatment with 2 g myo-inositol and 0.2 mg folic acid, a part of them are resistant and do not ovulate.

These non-responders to myo-inositol alone undergo the second phase of the study, receiving 2g myo-inositol and 0.2 mg folic acid plus 50 mg α-lactalbumin for three months. After this combined treatment, the majority of them ovulate, showing a hormone and lipid profile improvement. In addition, myo-inositol plasma levels at the end of the treatment are significantly higher than at baseline and comparable to those patients who respond positively to myo-inositol alone.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by PCOS according to Rotterdam ESHRE-ASRM criteria, with anovulation and infertility > 1 year

Exclusion Criteria:

* presence of other conditions causing ovulatory dysfunction, such as hyperprolactinemia or hypothyroidism, or androgen excess, such as adrenal hyperplasia or Cushing's syndrome, and also in the case of intake of other drugs that can potentially influence the ovulation.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Restoration of ovulation | after three months of treatment
  Ovulation was assessed using ultrasound examination on days 12, 14 and 20 of the cycle.

SECONDARY OUTCOMES:
Increase of myo-inositol plasma levels after the treatment with myo-inositol plus alpha-lactalbumin compared to the levels at the baseline | after three months of treatment
  Myo-inositol was dosed in plasma by means of gas chromatography-mass spectrometry

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Woman Health and Reproductive Medicine of Santo Spirito Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Montanino Oliva M, Buonomo G, Calcagno M, Unfer V. Effects of myo-inositol plus alpha-lactalbumin in myo-inositol-resistant PCOS women. J Ovarian Res. 2018 May 10;11(1):38. doi: 10.1186/s13048-018-0411-2. PMID 29747700